CLINICAL TRIAL: NCT01344434
Title: Angiographic CT of Renal Transplantation Candidate - Study
Brief Title: ACToR-study : Angiographic CT of Renal Transplantation Candidate - Study
Acronym: ACToR
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: M-20100270
Record Dates: First submitted 2011-04-08; First posted 2011-04-29 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-02

CONDITIONS: Renal Transplant Candidate for Right Kidney; Renal Transplant Candidate for Left Kidney

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study hypothesizes that renal transplantation candidates are diagnosed with significant Coronary Artery Disease (CAD) equal with non-invasive modalities as with invasive modalities. Therefore the investigators are investigating the ability of coronary computed tomographic angiography (cCTA), myocardial perfusion scintigraphy (MPS), acoustic CAD Patch and combination hereof to detect CAD as defined by invasive Coronary angiography (CAG).

DETAILED DESCRIPTION:
Chronic kidney disease is a known risk factor for cardiovascular disease and cardiovascular disease is the leading cause of mortality in end-stage renal disease (ESRD) patients. After renal transplantation one-half of all deaths are cardiac, usually in the first 5 years in the presence of a functional graft. Because of this renal transplantation candidates are undergoing cardiac pre-transplant risk stratification.

There is no consensus regarding which modality should be use for detection of CAD in this cardiac pre-transplant risk stratification. CAG is known as gold standard but is a invasive procedure with risk of complication.

The investigators wish to investigate the ability of detecting CAD as defined by invasive Coronary angiography (CAG) by clinical examination, blood test and non-invasive test (cCTA, MPS and acoustic CAD Patch). The investigators hypothesize that a single modality or combination of these with high sensitivity and specificity could diagnose significant CAD without the need of further invasive procedures.

This study will include 150 renal transplantations candidate.

ELIGIBILITY:
Inclusion Criteria:

* Endstage renal disease
* Preparing for renal transplantation
* Indication for CAG

Exclusion Criteria:

* Known allergy to iodinated contrast
* Women who are pregnant or nursing
* Severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease (CKD) who are renal transplantation candidates. Aged > 18
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To investigate the ability of non-invasive tests to detect CAD as defined by invasive angiography in renal transplantation candidates. | 2013 october
  Baseline results of coronary computed tomographic angiography (cCTA), myocardial perfusion scintigraphy (MPS), acoustic CAD Patch and combination hereof to detect CAD as defined by invasive Coronary angiography (CAG).

SECONDARY OUTCOMES:
To investigate the risk of Contrast-Induced Nephropathy (CIN) after cCTA and CAG. | 2013 october
  Blood sample of creatinine after contrast exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Winther, MD, Principal Investigator — Department of Cardiology, Skejby Sygehus, Denmark
Locations (1):
- Skejby Sygehus, Aarhus, Denmark

REFERENCES:
- [Derived] Dahl JN, Nielsen MB, Rasmussen LD, Ivarsen P, Williams MC, Svensson MHS, Birn H, Bottcher M, Winther S. Coronary Plaque Characteristics in Patients With Chronic Kidney Failure: Impact on Cardiovascular Events and Mortality. Circ Cardiovasc Imaging. 2024 Oct;17(10):e017066. doi: 10.1161/CIRCIMAGING.124.017066. Epub 2024 Sep 30. PMID 39344509
- [Derived] Winther S, Svensson M, Jorgensen HS, Rasmussen LD, Holm NR, Gormsen LC, Bouchelouche K, Botker HE, Ivarsen P, Bottcher M. Prognostic Value of Risk Factors, Calcium Score, Coronary CTA, Myocardial Perfusion Imaging, and Invasive Coronary Angiography in Kidney Transplantation Candidates. JACC Cardiovasc Imaging. 2018 Jun;11(6):842-854. doi: 10.1016/j.jcmg.2017.07.012. Epub 2017 Sep 13. PMID 28917674
- [Derived] Jorgensen HS, Winther S, Bottcher M, Hauge EM, Rejnmark L, Svensson M, Ivarsen P. Bone turnover markers are associated with bone density, but not with fracture in end stage kidney disease: a cross-sectional study. BMC Nephrol. 2017 Sep 6;18(1):284. doi: 10.1186/s12882-017-0692-5. PMID 28874132
- [Derived] Winther S, Bottcher M, Jorgensen HS, Bouchelouche K, Gormsen LC, Oczachowska-Kulik AE, Holm NR, Botker HE, Ivarsen PR, Svensson M. Coronary Calcium Score May Replace Cardiovascular Risk Factors as Primary Risk Stratification Tool Before Kidney Transplantation. Transplantation. 2016 Oct;100(10):2177-87. doi: 10.1097/TP.0000000000000992. PMID 26555948
- [Derived] Winther S, Svensson M, Jorgensen HS, Bouchelouche K, Gormsen LC, Pedersen BB, Holm NR, Botker HE, Ivarsen P, Bottcher M. Diagnostic Performance of Coronary CT Angiography and Myocardial Perfusion Imaging in Kidney Transplantation Candidates. JACC Cardiovasc Imaging. 2015 May;8(5):553-562. doi: 10.1016/j.jcmg.2014.12.028. Epub 2015 Apr 10. PMID 25869350